CLINICAL TRIAL: NCT05018143
Title: Suicide Prevention Intervention for Vulnerable Emerging Adult Sexual Minorities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jose Bauermeister, Chair, Department of Family & Community Health, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 849500
Record Dates: First submitted 2021-08-11; First posted 2021-08-24 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Suicide
Keywords: Sexual minority; Suicide; Emerging adults
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: The investigators will adapt a life skills intervention to increase the desire to live and reduce suicide ideation among at-risk emerging adult sexual minorities (EASM). STARS will embed components of the Safety Plan Intervention and modules to promote coping with discrimination, social support, and positive affect. We will pilot test STARS in a racially/ethnically diverse sample of 60 EASM who report past-month suicidal ideation. Eligible participants will provide informed consent and complete a Safety Planning Intervention with a licensed clinician. They then will be randomized to the control condition ("CC", n = 30) or STARS (n = 30). The investigators will follow participants for 6 months, with evaluations at 2, 4, and 6 months. Primary outcomes will be preliminary efficacy outcomes of suicidal ideation and behavior and hypothesized mechanisms of change (improved coping with discrimination, social support, positive affect) to estimate critical parameters for a future trial.
Who Masked: Outcomes Assessor
Masking Description: Outcomes evaluator will be blinded to randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STARS (Experimental): The investigators will deliver an online intervention focused on safety planning (STARS). The intervention content includes life skills interactive modules across 14 domains, a goal tracker, referral to community resources, and scheduling of peer mentoring sessions.
  Interventions: Behavioral: STARS
- Control Condition (Active Comparator): The investigators will deliver an in-person therapeutic session where participants can develop an individualized safety plan for use during a suicidal crisis, focusing on adaptive coping, addressing barriers or ambivalence, and strengthening their self-efficacy.
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: STARS — This intervention will use an online mobile application for teach life skills, coupled with peer mentoring to support the use of safety planning.
  Arms: STARS
Behavioral: Control condition — In this intervention, participants will receive the safety planning intervention.
  Arms: Control Condition

SUMMARY:
Emerging adult sexual minorities (EASM) are vulnerable to stressors that increase risk for suicidal ideation and behaviors. The investigators will examine a mobile application that leverages skills coaching and peer mentoring to reduce suicide risk for EASM. The online life skills intervention (iREACH) was developed to reduce a variety of negative health outcomes using telehealth with peer mentors. In Supporting Transitions to Adulthood and Reducing Suicide (STARS), investigators' interdisciplinary team will adapt iREACH to reduce suicidal ideation and behaviors among EASM. Then, investigators will pilot test STARS using in a racially/ethnically diverse sample of EASM with suicidal ideation. Participants will be randomized to receive an in-person brief, evidence-based safety planning protocol or to receive safety planning plus access to STARS. This project will identify the potential clinical utility of STARS for suicide prevention in a vulnerable, marginalized, population to inform a future larger efficacy RCT.

DETAILED DESCRIPTION:
Investigators will use the ADAPT-ITT framework to adapt a life skills intervention to increase the desire to live and reduce suicide ideation among at-risk emerging adult sexual minorities. STARS will embed components of the Safety Plan Intervention as well as modules focused on promoting coping with discrimination, social support, and positive affect. Investigators will pilot test STARS using a Type 1 Effectiveness-Implementation Hybrid Design in a racially/ethnically diverse sample of 60 EASM who report past-month suicidal ideation. Investigators will recruit EASM through social media advertising and invite them to an in-person screening. Eligible participants will provide informed consent and complete a Safety Planning Intervention with a licensed clinician, given the high-risk nature of the sample. They then will be randomized to the control condition ("CC", n = 30) or STARS (n = 30). Participants will be assessed at 2, 4, and 6 months. Primary outcomes will be preliminary efficacy outcomes of suicidal ideation and behavior and hypothesized mechanisms of change (improved coping with discrimination, social support, positive affect) to estimate critical parameters for a future trial. Secondary outcomes will be RE-AIM framework indicators (reach, adoption, implementation, maintenance). Our aims are: Aim 1: To conduct a systematic suicide prevention adaptation of a life skills intervention (STARS) that incorporates safety planning content and targets coping, social support, and positive affect using the ADAPT-ITT framework. Aim 2: To examine preliminary efficacy (suicidal ideation and behaviors) and mechanisms of action of STARS, relative to our control condition (safety planning protocol alone), using a prospective RCT design. Aim 3: Using RE-AIM metrics, to examine whether STARS has preliminary evidence for impacting intervention implementation outcomes among EASM compared to the control arm.

ELIGIBILITY:
Inclusion Criteria:

1. Identifies as a sexual minority
2. Lives in the Philadelphia Metropolitan Area;
3. Report suicide ideation in the prior month as verified in clinical interview;
4. Is aged 18-24 years (inclusive)
5. Daily use of a smartphone
6. Does not plan to move out of the region for the next 6 months
7. Consents to the study procedures

Exclusion Criteria:

1. Does not live in the Philadelphia Metropolitan Area;
2. Does not meet clinical criteria for suicide ideation in the prior month;
3. Is not between the ages of 18-24 years (inclusive)
4. Does not own a smartphone
5. Plan to move out of the region for the next 6 months
6. Does not consent to study procedures
7. Meets criteria for an unmanaged psychotic disorder

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José A Bauermeister, PhD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Center for the Treatment and Study of Anxiety, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be shared with the NIMH Data Archive.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The investigators will upload initial data 6 months after the onset of data collection with regular additions approximately every 6 months.
URL: https://nda.nih.gov/

REFERENCES:
- [Derived] Tran JT, Webster J, Wolfe JR, Ben Nathan J, Mayinja L, Kautz M, Oquendo MA, Brown GK, Mandell D, Mowery D, Bauermeister JA, Brown LA. Experiences of Peer Mentoring Sexual and Gender Minority Emerging Adults Who Are at Risk for Suicide: Mixed Methods Study. JMIR Form Res. 2025 Jan 29;9:e67814. doi: 10.2196/67814. PMID 39879591
- [Derived] Brown LA, Webster JL, Tran JT, Wolfe JR, Golinkoff J, Patel E, Arcomano AC, Ben Nathan J, Azat O'Connor A, Zhu Y, Oquendo M, Brown GK, Mandell D, Mowery D, Bauermeister JA. A Suicide Prevention Intervention for Emerging Adult Sexual and Gender Minority Groups: Protocol for a Pilot Hybrid Effectiveness Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 29;12:e48177. doi: 10.2196/48177. PMID 37773618
- Available data/document: Individual Participant Data Set: GUID — https://nda.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred through a targeted social media campaign.
Pre-assignment Details: Participants complete the safety planning intervention prior to randomization.
Period: Overall Study
Arm/Group | STARS | Control Condition
Started | 32 | 32
Completed | 27 (330: Completed all PM sessions and 2-4-and 6-month interviews but surveys were incomplete 118: Completed all PM sessions and 2-4-month assessments, but 6-month only completed the interview and not the survey 230: Completed first PM session and no follow-ups 250: Completed first PM session and no follow-ups 333: Completed first PM session and no follow-ups) | 27 (289: Lost to follow-up 329: 2 month completed, 4 and 6-months only completed interview, no survey 465: 2 and 4-months completed, 6 month completed interview only and no survey 569: 2 and 4-months completed, 6 month completed interview only and no survey 191: Withdrew participation at 2 month follow-up and completed interview only at this point, withdrew due to time commitment)
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants with past month suicidal ideation
Groups:
- Total: Total of all reporting groups
Arm/Group | STARS | Control Condition | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 64
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Mean] | 21 (1.983) | 21.8125 (1.595) | 21.40 (1.83)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant in the intervention arm identified as third-gender. Two participants did not report their sex assigned at birth.
  Participants
    number analyzed (Participants) | 29 | 32 | 61
    Female | 21 | 27 | 48
    Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 29 | 26 | 55
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 9 | 11 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 18 | 15 | 33
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Suicidal Ideation and Behavior
Description: The Columbia-Suicide Severity Rating Scale is an interview-rated measure that will be completed by a blind independent evaluator. The Columbia-Suicide Severity Rating Scale includes a measure of suicidal ideation (range 0-5: higher scores indicate more severe ideation). The measure has strong psychometric properties, including inter-rater reliability and internal consistency. The suicidal behavior and the suicidal ideation subscales have been shown to predict future suicidal behavior.
Time Frame: Change from baseline to 6 months
Population: Participants with past month suicidal ideation
Measure: Mean (Standard Deviation); unit: Mean Units on the CSSRS SI scale
Arm/Group | STARS | Control Condition
Number analyzed (Participants) | 32 | 32
Mean Units on the CSSRS SI scale
  Baseline | 2.625 (.870669) | 2.34375 (1.180743)
  2 months: number analyzed (Participants) | 29 | 31
  2 months | 1.37931 (1.115277) | 1.064516 (.9286364)
  4 months: number analyzed (Participants) | 29 | 30
  4 months | 1.37931 (1.2653) | .8333333 (1.147211)
  6 months: number analyzed (Participants) | 29 | 29
  6 months | 1.000 (1.101946) | 1.103448 (1.31868)

2. Secondary Outcome: Social Support
Description: Support from family respectively, will be measured through the Procidano and Heller Perceived Social Support from Family Scale. This five-item emotional support scale is rated on a 5-point scale (1=Not True; 5=Very True), where higher scores indicate greater social support. The measure has strong convergent and divergent validity, as well a strong test-retest reliability and internal consistency.
Time Frame: Change from baseline to 6 months
Population: Participants with past month suicidal ideation
Measure: Mean (Standard Deviation); unit: Mean score on family support
Arm/Group | STARS | Control Condition
Number analyzed (Participants) | 32 | 32
Mean score on family support
  Baseline | 3.42 (1.14) | 3.36 (1.27)
  2 months: number analyzed (Participants) | 28 | 29
  2 months | 3.61 (0.96) | 3.43 (1.20)
  4 months: number analyzed (Participants) | 29 | 27
  4 months | 3.34 (0.86) | 3.2 (0.92)
  6 months: number analyzed (Participants) | 24 | 25
  6 months | 3.45 (0.96) | 3.23 (1.19)

3. Secondary Outcome: Number of Participants Who Used Their Safety Plant at Least 1 Time
Description: Self-reported use of their safety plan
Time Frame: Every 2 months until 6 months
Population: Participants with past month suicidal ideation
Measure: Count of Participants; unit: Participants
Arm/Group | STARS | Control Condition
Number analyzed (Participants) | 32 | 32
Participants
  2 months: number analyzed (Participants) | 28 | 27
  2 months | 22 | 18
  4 months: number analyzed (Participants) | 27 | 28
  4 months | 20 | 18
  6 months: number analyzed (Participants) | 27 | 25
  6 months | 14 | 11

4. Secondary Outcome: Beck Scale for Suicide Ideation
Description: Sum of self-reported suicide ideation, with a possible range from 0 - 38, with higher values reflecting greater severity of suicidal ideation.
Time Frame: Change from baseline to 6 months
Population: Participants with past month suicidal ideation
Measure: Mean (Standard Deviation); unit: Score on the scale
Arm/Group | STARS | Control Condition
Number analyzed (Participants) | 32 | 32
Score on the scale
  Baseline | 7.41 (6.30) | 7.56 (7.41)
  2 months: number analyzed (Participants) | 28 | 30
  2 months | 5.79 (5.79) | 6.10 (6.96)
  4 months: number analyzed (Participants) | 23 | 27
  4 months | 5.48 (5.70) | 5.15 (5.68)
  6 months: number analyzed (Participants) | 27 | 26
  6 months | 4.15 (5.48) | 5.88 (7.20)

ADVERSE EVENTS:
Time Frame: 6 months
Description: N/A, Systematic assessment using the C-SSRS
Arm/Group | STARS | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT05018143/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT05018143/ICF_001.pdf